CLINICAL TRIAL: NCT01611779
Title: Functional Advancement and Suspension of the Tongue (FAST) as a Treatment for Obstructive Sleep Apnea
Brief Title: FAST as a Treatment for Obstructive Sleep Apnea
Acronym: FAST
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Slow enrollment
Sponsor: Siesta Medical, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011
Record Dates: First submitted 2012-05-29; First posted 2012-06-05 (Estimated); Results first posted 2017-01-06 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2017-01

CONDITIONS: Obstructive Sleep Apnea
Keywords: obstructive sleep apnea; tongue suspension
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Tongue suspension (Experimental): Tongue-based suspension
  Interventions: Device: Encore Tongue Suspension System

INTERVENTIONS:
Device: Encore Tongue Suspension System — The primary components of the Encore Tongue Suspension System consist of a suture passer, suspension line and bone screw.
  Other Names: Tongue suspension; FG0002

SUMMARY:
The objective of this study is to assess the feasibility and safety of tongue suspension using the Siesta Medical Encore Tongue Suspension System for the treatment of obstructive sleep apnea (OSA).

DETAILED DESCRIPTION:
Obstructive sleep apnea (OSA) has become a major health problem in the United States. With prevalence in middle-aged adults of 2-4% of the population, untreated OSA has been implicated in increased risk for cardiovascular disease, including hypertension and heart failure.

The first and most common treatment for OSA is continuous positive airway pressure (CPAP) treatment, utilized by an estimated 3 million Americans. CPAP is effective in reducing apnea-hypopnea index (AHI) is used properly. However, the nasal mask required for CPAP during sleep leads to poor acceptance and compliance rates. Published studies on CPAP have shown that only 58-8-% of patient accept CPAP therapy and further 65-90% of these patients exhibit long-term compliance with CPAP.

It is widely accepted that the region behind the tongue is a major site of collapse during obstructive sleep apnea. In fact there are many surgical procedures performed currently to address tongue based collapse. These include RF ablation of the tongue base, genioglossus advancement, hyoid suspension, maxillomandibular advancement, and tongue base suspension.

The current study is designed to evaluate the feasibility of tongue stabilization, and assess safety and treatment of the tongue stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Documented diagnosis of moderate obstructive sleep apnea (AHI 5-30/hour) measured within 12 months prior to the planned procedure
* Age >/= 20 and >/= 65
* Body Mass Index ,/= 32 (kg/m^2)
* Patient offered CPAP and has refused of failed to continue CPAP treatment or is not compliant with CPAP
* Signed informed consent to participate in this study

Exclusion Criteria:

* Prior OSA surgery
* Active systemic infection
* Allergy to any medication used during implantation
* Previous history of neck or upper respiratory tract
* Significant dysphagia or speech disorder

Anatomical

* Identified obvious palatal stenosis
* Enlarged tonsils (3+)
* Anatomy unable to accommodate the implant

Other

* Other medical, social, or psychological problems that , in the opinion of the investigator, precludes the patient from receiving this treatment and the procedures and evaluations pre- and post-treatment
* Enrollment in another pharmacological or medical device study that may effect or bias the results of this clinical study
* Unable and/or not willing to comply with treatment follow-up requirements
* Pregnancy (Female subjects of childbearing potential must have a negative pregnancy test prior to enrollment

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2012-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Goldberg, MD, Study Director — University of California, San Francisco
Locations (1):
- The Atlanta Snoring and Sleep Disorders Institute, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tongue Suspension
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients with obstructive sleep apnea were enrolled in the trial. Subjects meeting the inclusion and exclusion criteria were invited to participate in the trial. Subjects were treated with the the Encore System, and followed at 1 week, and then at 1, 3, and 12 months.
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 0
Gender [Count of Participants; unit: Participants]
  Female | 1
  Male | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 26.98 (3.78)
Prior OSA Surgery [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Place the Implant and Stabilize the Tongue
Description: Ability to place the implant and stabilize the tongue
Time Frame: Up to 7 weeks after the procedure
Measure: Count of Participants; unit: Participants
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 5
Participants | 5

2. Primary Outcome: Number of Participants Experiencing Complications
Description: Patient will be examined by the investigator at each of the follow-up visits for the presence of any untoward or unintended response to the device.
Time Frame: 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 5
Participants
  Headache | 1
  No Complications | 4

3. Secondary Outcome: Apnea Hypopnea Index
Description: 0 to >30/hour (high value represents worse outcome)
Time Frame: Baseline, 3, and 12 months
Population: Three (3) of 5 subjects returned for 3 month follow-up and 2 of 5 subjects returned for the 12 month follow-up.
Measure: Mean (Standard Deviation); unit: events/hour
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 5
events/hour
  Baseline | 24.2 (10.3)
  3 months: number analyzed (Participants) | 3
  3 months | 15.9 (7.8)
  12 months: number analyzed (Participants) | 2
  12 months | 34.6 (6.6)

4. Secondary Outcome: Functional Outcomes and Sleep Questionnaire (FOSQ)
Description: Questionnaire: 0 to 120 (high value represents better outcome)
Time Frame: Baseline, 1, 3, 12 months
Population: Four (4) of 5 total subjects had data at baseline and follow-up data.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 4
units on a scale
  Baseline | 17.2 (1.6)
  1 month | 18.2 (1.9)
  3 months | 18.1 (2.1)
  12 months | 17.2 (2.4)

5. Secondary Outcome: Snoring Scale (VAS)
Description: 0 to 10 (high value represents worse outcome)
Time Frame: Baseline, 1 week; 1 month, 3 months, 12 months
Population: Four (4) of 5 total subjects had data at baseline. Four (4) of 5 subjects had follow-up data at 1 week, 4 had follow-up data at 1 month, 3 had follow-up data at 3 months, and 2 had follow-up data at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 4
units on a scale
  Baseline | 5.5 (3.4)
  1 week | 2.6 (2.3)
  1 month | 1.8 (1.0)
  3 months: number analyzed (Participants) | 3
  3 months | 1.8 (1.6)
  12 months: number analyzed (Participants) | 2
  12 months | 1.7 (2.4)

6. Secondary Outcome: Epworth Sleeping Scale (ESS)
Description: 0 to 24 (high value represents worse outcome)
Time Frame: Baseline, 1, 3, 12 months
Population: Five (5) of 5 total subjects had data at baseline. Four (4) of 5 subjects had follow-up data at 1 week, 4 had follow-up data at 1 month, 4 had follow-up data at 3 months, and 2 had follow-up data at 12 months.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Tongue Suspension
Number analyzed (Participants) | 5
units on a scale
  Baseline | 12.4 (4.0)
  1 month: number analyzed (Participants) | 4
  1 month | 7.7 (2.2)
  3 months: number analyzed (Participants) | 4
  3 months | 7 (2.4)
  12 months: number analyzed (Participants) | 2
  12 months | 6.5 (2.1)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Tongue Suspension
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 1/5
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tongue Suspension (N=5)
Headache (General disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No